CLINICAL TRIAL: NCT02085070
Title: A Phase 2 Study of MK-3475 in Patients With Metastatic Melanoma and Non-Small Cell Lung Cancer With Untreated Brain Metastases
Brief Title: MK-3475 in Melanoma and NSCLC Patients With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Harriet Kluger, Associate Professor, Internal Medicine, Oncology, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1401013290; IND 121564 (Other: FDA)
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-02

CONDITIONS: Melanoma; Non-Small Cell Lung Cancer; Brain Metastases
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melanoma patients (Experimental): After establishing eligibility criteria, for patients with melanoma the investigator will determine at least one lesion that requires local therapy (surgical resection or LITT) based on size, location, and/or risk of hemorrhage; this will be considered the "surgical lesion". All other eligible brain lesions will be considered "clinically evaluable lesions" and will be followed by modified RECIST (mRECIST) criteria to determine best response.
  Interventions: Drug: MK-3475
- Non-small cell lung cancer patients (Other): NSCLC patients are not required to have a "surgical lesion" but must have at least one "clinically evaluable lesion" in the central nervous system. Patients on NSCLC are required to have formalin-fixed, paraffin-embedded tumor tissue available for biomarker analysis.
  Interventions: Drug: MK-3475

INTERVENTIONS:
Drug: MK-3475 — IV MK-3475

SUMMARY:
The purpose of this trial is to study the activity of MK-3475 in untreated brain metastases from melanoma or non-small cell lung cancer.

DETAILED DESCRIPTION:
While recent advances in the treatment of metastatic melanoma and NSCLC (non-small cell lung cancer) with agents targeting PD-1 are striking, there remains a significant need to develop therapies for patients with untreated brain metastases who were excluded from prior trials with MK-3475 and the majority of other studies in these diseases. The brain is a common site of disease spread in many solid tumors, most notably metastatic melanoma and NSCLC. 10-40% of patients with metastatic melanoma develop brain metastases during their lifetime and >75% have brain metastases at autopsy. Overall, historical melanoma patient cohorts have reported a median survival of patients with brain metastases in the order of 2.5 - 4 months despite use of whole brain radiation therapy (WBRT) and surgery. One older patient series showed a median survival of < 4 months in melanoma patients with brain metastases and a neurological death rate of >30% despite the treatment of intracranial metastases with whole brain radiation therapy (WBRT). Among those with NSCLC, 10% have brain metastases at presentation and another 30% develop them over the course of their disease. Survival after the development of brain metastases is as dismal in those with NSCLC as it is for melanoma. Multifocal disease is common in both of these diseases, with about half of patients with CNS disease presenting with more than one brain lesion.

Patients with untreated brain metastases have been excluded from most clinical trials of systemic therapy for two reasons: (1) historically their prognosis has been poor (overall survival ≤ 4 months) and (2) experimental drugs are presumed to not penetrate the blood brain barrier (BBB) or BBB penetration is not well studied. In melanoma, for example, one phase III study evaluating ipilimumab excluded patients with untreated brain metastases and another study evaluating ipilimumab and dacarbazine excluded all patients with a history of brain metastases, regardless of prior treatment. A subsequent trial with ipilimumab for patients with untreated brain metastases indeed showed that the drug had some activity in treating CNS disease. In the initial vemurafenib studies, patients with progressing or unstable CNS metastases were excluded. The pivotal BRIM-3 trial excluded patients with brain metastases unless metastases had been definitively treated more than three months prior to trial enrollment. Both temodar and sorafenib cross the BBB. Initial studies with sorafenib alone and in combination with chemotherapy excluded patients with active brain metastases. A combination study of temodar and sorafenib in patients with or without brain metastases showed modest activity in patients without a history of prior temodar, and was thought to be favorable in part due to local therapies. Although a number of studies have been conducted for melanoma patients with untreated brain metastases using established therapies, most initial clinical trials with novel agents exclude these patients. A recent trial with dabrafenib, an inhibitor of mutated B-raf, is an exception to the long-standing paradigm. A phase I/II study of this agent included a subset of patients with untreated brain metastases. At the 2010 meeting of the European Society for Medical Oncology, Long et al reported that nine of the ten patients with untreated cerebral metastases enrolled in this trial had shrinkage of their brain lesions. This was the basis for a recent phase II trial of dabrafenib specific for patients with untreated brain metastases61. In NSCLC, a small number of trials have shown that combination chemotherapy regimens can induce a response in the CNS with untreated brain metastases with a median PFS up to 4 months. These studies demonstrate that asymptomatic brain metastases, similar to asymptomatic metastases in other sites, can be treated systemically on clinical trials, and that drug activity in the CNS is not necessarily different than in other metastatic locations.

Current standard of care for brain metastases that require immediate local intervention (based on symptoms, location, size, or other concerning features) is craniotomy with resection or radiation therapy. As an adjunct to standard craniotomy, LITT is emerging as a new, minimally invasive local therapy to treat previously surgically inaccessible brain metastases. Not only is cell death instantaneous, thus decreasing the risk of delayed intra-tumoral hemorrhage, but another theoretical advantage of using LITT as part of management of brain metastases is that the hyperthermia breaks down the blood brain barrier at the edge of the coagulation region thereby possibly increasing access of chemotherapeutic agents into the lesion. In patients in whom either craniotomy or LITT are performed, biopsies of tumor and surrounding normal brain can also be obtained at the time of local therapy.

The purpose of this trial is to study the activity of MK-3475 in untreated brain metastases from melanoma or NSCLC. Given the promising initial results of MK-3475 in these diseases but the lack of data in patients with untreated brain metastases thus far, this trial will study treatment in this patient population. Additionally, for patients with melanoma this trial requires local therapy with craniotomy or LITT to at least 1 brain lesion prior to systemic therapy, thereby allowing the acquisition of brain tumor tissue for correlative studies on biomarkers that may be predictive of clinical response in the CNS and systemically. There will also be a biopsy of an extra-cerebral metastasis when feasible, particularly when tissue from the brain lesion is not obtained in patients with NSCLC.

Upon results entry, the primary outcome measure was aligned as originally presented in the study protocol (attached with results).

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven metastatic melanoma or NSCLC as follows:

   1. Patients with metastatic melanoma must have untreated brain metastases including:

      * At least one cerebral metastasis that requires local intervention and is amenable to craniotomy or LITT therapy either due to symptoms, lesion size, location, edema or hemorrhage ("surgical lesion"). Alternatively, a patient may be eligible if a cerebral metastasis was resected or biopsied any time prior to enrollment and there is tumor tissue available for analysis.
      * At least one cerebral metastasis that is at least 5 mm AND twice the MRI slice thickness, but less than 20 mm, that is asymptomatic and does not require local therapy at the time of enrollment ("clinically evaluable lesion(s)"). OR
   2. Patients with stage IV NSCLC with at least one cerebral metastasis that is at least 5 mm AND twice the MRI slice thickness, but less than 20 mm, that is asymptomatic and does not require local therapy at the time of enrollment ("clinically evaluable lesion(s)").
2. Age ≥18
3. ECOG performance status < 2
4. Any number of previous treatments with the exception of previous inhibitors of PD-1, PD-L1, or PD-L2; other prior systemic therapies must have been administered at least 2 weeks before administration of MK-3475 with the exception of bevacizumab which must have been administered at least 4 weeks prior to MK-3475. Patients are not required to have had prior systemic therapy. The exception to this is patients with NSCLC who test negative for PD-L1 expression or are unevaluable for PD-L1 expression must have received prior platinum-based chemotherapy for entry into Cohort 2. Note: Ipilimumab treatment should have been administered at least 4 weeks prior to the start of MK-3475.
5. Life expectancy of at least 3 months
6. A history of previously treated brain metastases is allowed, provided that at least 14 days have lapsed between radiation and initiation of MK-3475. Any lesion present at the time of WBRT or included in the stereotactic radiotherapy field (or within 2mm of the treated lesion) will NOT be considered evaluable unless it is new or documented to have progressed since treatment.
7. PD-L1 expression in tumor tissue from any site is required for patients with NSCLC for entry into Cohort 1. Tumor tissue must be obtained after the last systemic therapy. PD-L1 expression will be analyzed by a Merck assay. For NSCLC Cohort 2, patients may test PD-L1 negative or may be unevaluable for PD-L1 expression (i.e. insufficient tumor tissue). PD-L1 expression is not required for patients with melanoma, but melanoma patients are required to submit an extra-cerebral specimen for analysis, unless it is not feasible to obtain one.
8. Patients must have normal organ and marrow function as defined per protocol.
9. For women of childbearing potential, agreement to the use of two acceptable methods of contraception, including one barrier method, during the study and for 6 months after discontinuation of MK-3475.
10. For men with female partners of childbearing potential, agreement to use a latex condom, and to advise their female partner to use an additional method of contraception during the study and for 6 months after discontinuation of MK-3475.
11. Negative serum or urine pregnancy test within 72 hours of commencement of treatment in premenopausal women.
12. Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Symptomatic brain metastases. Symptoms may be present from the surgical lesion prior to resection or LITT but must have resolved by the time of administration of study drug.
2. Patients with brain metastases for whom complete surgical resection is clinically appropriate.
3. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy to the lung or brain within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Previous radiation to other sites may be completed at any time prior to initiation of MK-3475.

   1. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
   2. Note: Toxicity that has not recovered to ≤ Grade 1 is allowed if it meets the inclusion requirements for laboratory parameters.
4. Has had prior treatment with any other anti-PD-1 or PD-L1 or PD-L2 agent or an antibody targeting other immune-regulatory receptors or mechanisms. Examples of such antibodies include (but are not limited to) antibodies against IDO, PD-L1, IL-2R, GITR. Prior ipilimumab, IL2, bevacizumab and adoptive cell therapy is allowed.
5. The use of corticosteroids to control cerebral edema or treat neurologic symptoms will not be allowed, and patients who previously required corticosteroids for symptom control must be off steroids for at least 2 weeks. Low-dose steroid use (≤10 mg of prednisone or equivalent) as corticosteroid replacement therapy is allowed
6. Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Presence of leptomeningeal disease
8. Has an active automimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of inhaled steroids or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
9. Pregnancy or breast feeding. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MK-3475, breastfeeding must be discontinued if the mother is treated with MK-3475.
10. Patients may not be receiving any other investigational agents and may not have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
11. Either a concurrent condition (including medical illness, such as active infection requiring treatment with intravenous antibiotics or the presence of laboratory abnormalities) or history of a prior condition that places the patient at unacceptable risk if he/she were treated with the study drug or a medical condition that confounds the ability to interpret data from the study.
12. Concurrent, active malignancies in addition to those being studied (other than cutaneous squamous cell carcinoma or basal cell carcinoma)
13. Any contraindication to MRI (i.e. patients with pacemakers or other metal implanted medical devices). An MRI safety questionnaire is required prior to MR imaging.
14. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
15. Has a known Human Immunodeficiency Virus (HIV), Hepatitis B (HBV), or Hepatitis C (HCV) infection.
16. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
17. Evidence of interstitial lung disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-03; Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Kluger, MD, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Center at Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldberg SB, Schalper KA, Gettinger SN, Mahajan A, Herbst RS, Chiang AC, Lilenbaum R, Wilson FH, Omay SB, Yu JB, Jilaveanu L, Tran T, Pavlik K, Rowen E, Gerrish H, Komlo A, Gupta R, Wyatt H, Ribeiro M, Kluger Y, Zhou G, Wei W, Chiang VL, Kluger HM. Pembrolizumab for management of patients with NSCLC and brain metastases: long-term results and biomarker analysis from a non-randomised, open-label, phase 2 trial. Lancet Oncol. 2020 May;21(5):655-663. doi: 10.1016/S1470-2045(20)30111-X. Epub 2020 Apr 3. PMID 32251621
- [Background] Kluger HM, Chiang V, Mahajan A, Zito CR, Sznol M, Tran T, Weiss SA, Cohen JV, Yu J, Hegde U, Perrotti E, Anderson G, Ralabate A, Kluger Y, Wei W, Goldberg SB, Jilaveanu LB. Long-Term Survival of Patients With Melanoma With Active Brain Metastases Treated With Pembrolizumab on a Phase II Trial. J Clin Oncol. 2019 Jan 1;37(1):52-60. doi: 10.1200/JCO.18.00204. Epub 2018 Nov 8. PMID 30407895
- [Background] Goldberg SB, Gettinger SN, Mahajan A, Chiang AC, Herbst RS, Sznol M, Tsiouris AJ, Cohen J, Vortmeyer A, Jilaveanu L, Yu J, Hegde U, Speaker S, Madura M, Ralabate A, Rivera A, Rowen E, Gerrish H, Yao X, Chiang V, Kluger HM. Pembrolizumab for patients with melanoma or non-small-cell lung cancer and untreated brain metastases: early analysis of a non-randomised, open-label, phase 2 trial. Lancet Oncol. 2016 Jul;17(7):976-983. doi: 10.1016/S1470-2045(16)30053-5. Epub 2016 Jun 3. PMID 27267608
- [Derived] Qian JM, Yu JB, Mahajan A, Goldberg SB, Kluger HM, Chiang VLS. Frequent Use of Local Therapy Underscores Need for Multidisciplinary Care in the Management of Patients With Melanoma Brain Metastases Treated With PD-1 Inhibitors. Int J Radiat Oncol Biol Phys. 2019 Dec 1;105(5):1113-1118. doi: 10.1016/j.ijrobp.2019.08.053. Epub 2019 Aug 31. PMID 31479702
- [Derived] Qian JM, Mahajan A, Yu JB, Tsiouris AJ, Goldberg SB, Kluger HM, Chiang VLS. Comparing available criteria for measuring brain metastasis response to immunotherapy. J Neurooncol. 2017 May;132(3):479-485. doi: 10.1007/s11060-017-2398-8. Epub 2017 Mar 8. PMID 28275886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 NSCLC patients were ineligible based on PD-L1.
Pre-assignment Details: Patients were assigned to a cohort based on tumor type.
Period: Overall Study
Arm/Group | Melanoma Patients | Non-small Cell Lung Cancer Patients
Started | 23 | 42
Completed | 23 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melanoma Patients | Non-small Cell Lung Cancer Patients | Total
Number analyzed (Participants) | 23 | 42 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 27 | 37
  >=65 years | 13 | 15 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 28 | 36
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 23 | 36 | 59
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 23 | 35 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 23 | 42 | 65

OUTCOME MEASURES:

1. Primary Outcome: Overall Response in the Brain by mRECIST
Description: RECIST criteria v1.1 was modified to account for differences in measuring the response of clinically evaluable brain lesions as opposed to systemic lesions (modified RECIST, or mRECIST). Size was considered the tumor's largest diameter. Measurements from multiple lesions were summed to calculate the sum of the diameters (SD). The SD calculated on a baseline scan performed within 28 days of study drug initiation was used as a reference to determine the objective response of the clinically evaluable lesions.
  mRECIST differ from RECIST v1.0 in allowing lesions measuring 5mm or less for response evaluation, provided that the MRI slice thickness was no more than 2.5mm. Seeing that the primary trial endpoint was brain metastasis response, up to 5 lesions were used for evaluation.
  Complete response (CR) constitutes complete disappearance of all target lesions, partial response (PR) constitutes >= 30% decrease in the sum of the sum of the largest diameter of target
Time Frame: 8 weeks
Population: modified RECIST 1.1 was used to determine response
Measure: Number; unit: participants
Arm/Group | Melanoma Patients | Non-small Cell Lung Cancer Patients
Number analyzed (Participants) | 23 | 42
participants
  progression/stable | 17 | 31
  better response | 6 | 11
Statistical Analysis 1: Comparison: Non-small Cell Lung Cancer Patients; Each group was assessed individually. The primary goal of this study is to determine the efficacy of MK-3475 in patients with untreated brain metastases from NSCLC. The primary endpoint is the brain metastasis response rate (BMRR). A drug with minimal activity would be expected to have a BMRR of 10%; Test type: Superiority — A response of > 10% of patients was defined as superior; % response = 29.7, 95% CI 2-sided [15.9 to 47.0]
Statistical Analysis 2: Comparison: Melanoma Patients; Each group was assessed individually. The primary goal of this study is to determine the efficacy of MK-3475 in patients with untreated brain metastases from melanoma. The primary endpoint is the brain metastasis response rate (BMRR). A drug with minimal activity would be expected to have a BMRR of 10%; Test type: Superiority — A response of > 10% of patients was defined as superior; % of patients = 26.0, 95% CI 2-sided [10.0 to 48.0]

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Melanoma Patients | Non-small Cell Lung Cancer Patients
All-Cause Mortality (participants affected / at risk) | 16/23 | 35/42
Serious Adverse Events (participants affected / at risk) | 5/23 | 5/42
Other Adverse Events (participants affected / at risk) | 13/23 | 35/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melanoma Patients (N=23) | Non-small Cell Lung Cancer Patients (N=42)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Adrenal Insufficienvy (Endocrine disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melanoma Patients (N=23) | Non-small Cell Lung Cancer Patients (N=42)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (6)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 21 (30)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 14 (26)
Nausea (Gastrointestinal disorders) | 7 (7) | 12 (17)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (6)
Chills (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 13 (13) | 35 (65)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 18 (26)
Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (10)
Ataxia (Nervous system disorders) | 3 (3) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 2 (2)
Confusion (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 10 (13)
Dysphasia (Nervous system disorders) | 2 (2) | 0 (0)
Gait disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 15 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 26 (42)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (11)
Hypothyroidism (Endocrine disorders) | 1 (1) | 6 (8)
Floaters (Eye disorders) | 0 (0) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (4)
Edema limbs (General disorders) | 0 (0) | 10 (14)
Fever (General disorders) | 1 (1) | 3 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 5 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (4)
Creatinine increased (Investigations) | 0 (0) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 17 (25)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 13 (25)
Seizure (Nervous system disorders) | 1 (1) | 3 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 9 (11)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 7 (8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 21 (28)
Hypertension (Vascular disorders) | 0 (0) | 7 (8)
Thromboembolic event (Vascular disorders) | 0 (0) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT02085070/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT02085070/Prot_SAP_001.pdf